CLINICAL TRIAL: NCT04052555
Title: A Phase 1b Study of Berzosertib in Combination With Radiation Therapy to Overcome Therapeutic Resistance in Chemotherapy Resistant Triple Negative and Estrogen and/or Progesterone Receptor Positive, HER2 Negative Breast Cancer
Brief Title: Testing the Addition of an Anti-cancer Drug, Berzosertib, to the Usual Treatment (Radiation Therapy) for Chemotherapy-Resistant Triple-Negative and Estrogen and/or Progesterone Receptor Positive, HER2 Negative Breast Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2019-05187; NCI-2019-05187 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10291 (Other: Dana-Farber - Harvard Cancer Center LAO); 10291 (Other: CTEP); UM1CA186686 (NIH); UM1CA186709 (NIH)
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Bilateral Breast Carcinoma; HER2-Negative Breast Carcinoma; Localized Breast Carcinoma; Recurrent Breast Carcinoma; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — berzosertib; Specimen Handling; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (berzosertib, radiation therapy) (Experimental): Patients receive berzosertib IV over 60 minutes BIW for 5 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo RT 5 days a week for 5-6 weeks depending on the type of surgery undergone. Patients also undergo a collection of blood on study.
  Interventions: Drug: Berzosertib; Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Berzosertib — Given IV
  Other Names: 2-Pyrazinamine, 3-(3-(4-((Methylamino)methyl)phenyl)-5-isoxazolyl)-5-(4-((1-methylethyl)sulfonyl)phenyl)-; M 6620; M6620; VX 970; VX-970; VX970
Procedure: Biospecimen Collection — Correlative studies
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Radiation: Radiation Therapy — Undergo RT
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase Ib trial studies the best dose of berzosertib when given together with the usual treatment (radiation therapy) in treating patients with triple negative or estrogen receptor and/or progesterone receptor positive, HER-2 negative breast cancer. Berzosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy rays to kill tumor cells and shrink tumors. Giving M6620 and radiation therapy may kill tumor cells more effectively than radiation alone or shrink or stabilize breast cancer for longer than radiation therapy alone.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the recommended phase 2 dose of twice weekly berzosertib administered concurrently with conventionally fractionated radiation therapy (RT) to the breast/chest wall and regional nodes.

SECONDARY OBJECTIVES:

I. To describe the nature of toxicity that develops when an ATR inhibitor is administered concurrently with RT for breast cancer using provider assessments.

II. To assess long-term locoregional control, disease-free survival, distant disease-free survival, and overall survival of patients treated with this approach.

III. To explore symptomatic adverse events and tolerability of berzosertib being administered concurrently with RT using patient-reported outcomes (PROs).

IV. To assess for alterations in deoxyribonucleic acid (DNA) damage response and repair genes, including effectors and regulators of homologous recombination (HR), in pre-chemotherapy biopsy specimens and post-chemotherapy surgical resection specimens using whole exome sequencing (WES) and ribonucleic acid (RNA) sequencing (RNAseq), and to correlate HR deficiency with disease-free survival.

V. To identify somatic alterations in circulating cell-free DNA (cfDNA) at baseline, mid-treatment, end-of-treatment, and follow-up and to correlate cfDNA with disease-free survival.

EXPLORATORY OBJECTIVES:

I. To compare the baseline and post-treatment skin microbiome and make exploratory correlations with severe provider and patient-reported toxicity.

II. To explore dose-volume parameters associated with acute and late provider and patient-reported toxicity following berzosertib administration concurrent with RT.

III. To identify circulating tumor cell (CTC) positivity at baseline, mid-treatment, end-of-treatment, and follow-up and to correlate CTC positivity or the combination of CTC positivity and cfDNA with disease-free survival.

IV. To evaluate pre-treatment and post-treatment differential abundance of peripheral blood immune cell populations identified by cytometry by time-of flight (CyTOF).

V. To evaluate associations of the pre-treatment and post-treatment peripheral blood immune phenotype (as assessed by CyTOF) with disease-free survival, distant disease-free survival and overall survival.

VI. To explore the USP21-ATR pathway and its association with epithelial to mesenchymal transition (EMT) in therapeutically resistant breast cancer specimens at pre-treatment and post-treatment timepoints using immunohistochemistry (IHC) and RNAseq.

OUTLINE: This is a dose-escalation study of berzosertib.

Patients receive berzosertib intravenously (IV) over 60 minutes twice weekly (BIW) for 5 weeks in the absence of disease progression or unacceptable toxicity. Patients undergo RT 5 days a week for 5-6 weeks depending on the type of surgery undergone. Patients also undergo a collection of blood on study.

After completion of study treatment, patients are followed up weekly for 4 weeks, at 12 months, then yearly for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age >= 18 years. Note: Because no dosing or adverse event data are currently available on the use of berzosertib in combination with radiation therapy in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Patient with non-metastatic, histologically confirmed primary estrogen receptor (ER) =< 10%, progesterone receptor (PR) =< 10%, and HER2-negative breast cancer (triple negative breast cancer [TNBC]) either using the baseline biopsy specimen or the post-neoadjuvant chemotherapy (NAC) residual surgical specimen and RCB2 or RCB3, as defined by Symmans et al., 2007, and received neoadjuvant anthracycline and/or taxane-based chemotherapy OR Patient has non-metastatic, histologically confirmed primary ER > 10% and/or PR > 10%, HER2-negative breast cancer with RCB3 and received neoadjuvant anthracycline and/or taxane-based chemotherapy OR Patient has locoregionally recurrent TNBC or ER >10% and/or PR >10%, HER2-negative breast cancer.

  * Note: Results from any Clinical Laboratory Improvement Act (CLIA)-certified lab are acceptable for the purpose of determining study eligibility.
  * Note: For patients with primary breast cancer, there is no minimum number of neoadjuvant cycles required provided the patient received an anthracycline or taxane preoperatively. Patients with locoregionally recurrent breast cancer are not required to have received preoperative chemotherapy
* Patient has undergone total mastectomy or wide local excision with axillary staging, and the margins of the resected wide local excision or mastectomy specimens are free of invasive tumor and ductal carcinoma in situ (DCIS) or patient has undergone axillary surgery for regionally recurrent breast cancer. Unresected axillary level III, internal mammary, and supraclavicular nodal disease is permitted.

  * Note: For patients who have undergone mastectomy, immediate reconstruction is allowed
* Patients must have completed their final breast surgery, including re-excision of margins for invasive cancer and DCIS, within 90 but not fewer than 21 days prior to registration unless patient received postoperative chemotherapy in which case patients must have completed their adjuvant chemotherapy within 90 days but not fewer than 28 days prior to registration
* The patient must have recovered from surgery with the incision completely healed and no signs of infection prior to registration
* Patients must be proceeding with breast/chest wall and regional nodal irradiation including internal mammary node treatment. For patients with bilateral breast cancer, RT must be indicated and administered only to one side
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Willing to provide tissue and blood samples for correlative research
* Leukocytes >= institutional lower limit of normal (LLN)
* Absolute neutrophil count >= institutional LLN
* Platelets >= institutional LLN
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< 1.1 mg/dL OR
* Glomerular filtration rate (GFR) >= 45 mL/min/1.73 m^2 for patients with creatinine levels above 1.1 mg/dL
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Negative urine or serum pregnancy test for individuals of childbearing potential. Note: The effects of berzosertib on the developing human fetus are unknown. For this reason and because DNA-damage repair inhibitors as well as radiation used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation, and for 6 months after completion of berzosertib administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 6 months after completion of berzosertib administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy within 4 weeks prior to entering the study
* Prior RT to the ipsilateral chest wall or ipsilateral breast or thorax. Individuals with prior RT to the contralateral breast or chest wall are eligible
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia and grade 1-2 taxane-induced neuropathy which will be permitted
* Patients who are receiving any other investigational agents or concomitant anti-neoplastic treatment, except endocrine therapies and bisphosphonates which are permitted without restriction even during protocol treatment. Postoperative chemotherapy is allowed but must be discontinued >28 days prior to registration
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to berzosertib
* Berzosertib is primarily metabolized by CYP3A4; therefore, concomitant administration with strong inhibitors of CYP3A4 (e.g., ketoconazole, itraconazole, clarithromycin, ritonavir, indinavir, nelfinavir, and saquinavir) or inducers of CYP3A4 (e.g., rifampin, phenytoin, carbamazepine, phenobarbital, St. John's wort) should be avoided. Patients requiring any medications or substances that are strong inhibitors or inducers of CYP3A during the course of the study and for 14 days prior to enrollment are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness. This includes but is not limited to, ongoing uncontrolled serious infection requiring IV antibiotics at the time of registration, symptomatic congestive heart failure, unstable angina pectoris, symptomatic/uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Active systemic lupus, scleroderma, or dermatomyositis with a CPK level above normal
* Pregnant women are excluded from this study because berzosertib as a DNA damage repair inhibitor may have the potential for teratogenic or abortifacient. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with berzosertib, breastfeeding should be discontinued if the mother is treated with berzosertib
* Patients with known hereditary syndromes predisposing to radiosensitivity such as Li Fraumeni syndrome and ataxia telangiectasia are excluded from the study. Patients with mutations in breast cancer predisposition genes such as BRCA1, BRCA2, PALB2, CHEK2, and ATM are eligible
* Patients with a prior or concurrent malignancy, excluding non-melanoma skin cancers and non-invasive cancers whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2027-02-24 (Estimated); Study Completion 2027-02-24 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of berzosertib | Up to 4 weeks post treatment
  The maximum tolerated dose will be defined as the highest dose level with a dose-limiting toxicity rate closest to 0.25 and =< .33.

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 3 years
  Will be defined by the National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 and will be summarized descriptively for each dose level and the entire cohort. The number and severity of all AEs (overall and by dose-level) will be tabulated and summarized in this patient population. The grade 3+ AEs will also be described and summarized in a similar fashion.
Time to progression | From study registration until the tumor recurs in the ipsilateral breast, chest wall, axillary, supracavicular or internal mammary nodes (if before or synchronous with a systemic recurrence), assessed up to 3 years
  Locoregional control will be split by each dose level and analyzed descriptively using Kaplan-Meier methodology.
Disease-free survival (DFS) | From study registration until the tumor recurs or the patient dies, whichever comes first, assessed up to 3 years
  Will be split by each dose level and analyzed descriptively using Kaplan-Meier methodology.
Distant DFS | From study registration until distant disease recurs or the patient dies, whichever comes first, assessed up to 3 years
  Will be split by each dose level and analyzed descriptively using Kaplan-Meier methodology.
Overall survival | From study registration until death due to any cause, assessed up to 3 years
  Will be split by each dose level and analyzed descriptively using Kaplan-Meier methodology.
Change in patient-related outcomes (PRO) | Baseline up to 3 years
  Patient reported physical well-being, fatigue, skin toxicity (as measured by the PRO-CTCAE) and overall quality of life (as measured by the Breast-Q) will be summarized. The PRO-CTCAE data will be evaluated for data quality, to characterize baseline symptom status of patients on study and the change over time, to explore the development of symptomatic AEs and the change over time, and to explore the patient scores with other relevant clinical information, including clinician graded AEs. Changes in Breast-Q scores through time will be analyzed using graphical methods separately for each treatment level.
Alterations in deoxyribonucleic acid damage response and repair genes | Up to 3 years
  Will include effectors and regulators of homologous recombination (HR) and be correlated with HR deficiency with disease-free survival. Descriptive statistics (i.e., mean, median, standard deviation, and range) and graphical methods (i.e., boxplots, jitter plots) will be used to summarize and compare the relapses by different dose levels. The number of relapses between the HR-deficient versus (vs.) the HR-proficient patients will be compared using a Chi-square test or independence or Fisher's Exact test. DFS for the HR-deficient and HR-proficient patients will be analyzed using Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Mutter, Principal Investigator — Dana-Farber - Harvard Cancer Center LAO
Locations (14):
- United States (14):
  - Mayo Clinic Hospital in Arizona, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Texas Medical Branch, Galveston, Texas
  - Farmington Health Center, Farmington, Utah
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/55/NCT04052555/ICF_000.pdf